CLINICAL TRIAL: NCT05130346
Title: Effects of Mindfulness Based Stress Reduction Intervention in Patients With Non-alcoholic Fatty Liver Disease: Beyond the Paradigm of Weight Loss.
Brief Title: Effects of Mindfulness Based Stress Reduction Intervention in Patients With Non-alcoholic Fatty Liver Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is being withdrawn due to difficulties enrolling participants and the loss of the study coordinator
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20023471
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Fatty Liver, Nonalcoholic; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction (MBSR) (Experimental)
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR)
- Standard of Care (SOC) (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) — Participants will be asked to attend group meetings for mindfulness training. Each meeting will last approximately one hour and will take place online via Zoom. The meetings will occur on a weekly basis, over an 8-week period.
  Arms: Mindfulness Based Stress Reduction (MBSR)

SUMMARY:
The purpose of this research study is to find out about the usefulness of mindfulness for weight loss and improvement of physical and mental health in people who have non-alcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
Adding mindfulness to lifestyle changes for weight loss may improve fatty liver disease in particular and overall health and well-being in general by helping sustain weight loss and maintain a healthy lifestyle. This study will allow researchers to learn more about it.

Non-alcoholic fatty liver disease is a condition where there is accumulation of excess fat in the liver of people who drink little or no alcohol. It is part of the metabolic syndrome characterized by diabetes, or pre-diabetes (insulin resistance), being overweight or obese, elevated blood lipids, as well as high blood pressure, all are risk factors for the disease.

In this study, participants will receive usual care, and in addition, they may be asked to participate in a mindfulness-based stress reduction program for 8 weeks. Usual care involves the routine clinic follow up visits and routine lab tests and imaging studies.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of NAFLD and ALT >35 U/dl.
2. At least 2 features of Metabolic syndrome (defined by Adult Treatment Panel III (2005 revision)).
3. Age 18-80 years.
4. BMI ≥25 Kg/m2.
5. Capable of providing written or signed informed consent.

Exclusion Criteria:

1. Any known cause of liver disease other than NAFLD as confirmed by patient's history, laboratory data, and/or histological findings.
2. Decompensated liver cirrhosis based on laboratory data and clinical manifestations (varices, ascites, or encephalopathy).
3. Any previous experimental interventional treatment of NAFLD or NASH within the past 3 months.
4. Pre-existing diseases/conditions that could interfere with the results or the completion of this trial based on the investigator's judgment.
5. Unstable metabolic syndrome and other serious chronic medical conditions.
6. Unstable type 2 diabetes (any of the following):

   * Requiring medication adjustment within the last 3 months.
   * Patients requiring GLP-1 agonists treatment.
   * No more than 10% modification in insulin dose if on insulin.
   * If on SGLT-2 inhibitors, need to be on stable dose with more than 5% weight loss in the last 3 months.
7. Unable to adhere to out-patient clinic management program.
8. Do not speak English on a daily-user level.
9. Pregnant or planning to become pregnant within the following 6 months.
10. Active substance use disorder.
11. Does not accept follow-ups over 1 year from time of inclusion (T0).
12. Inmates.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in total body weight | Baseline to 6 months
  Relative change (%) in total body weight at 6 months (T1) from baseline (T0).
Change in bilirubin | Baseline to 6 months
  Relative change (%) in bilirubin at 6 months (T1) from baseline (T0).
Change in alanine transaminase (ALT) | Baseline to 6 months
  Relative change (%) in ALT at 6 months (T1) from baseline (T0).
Change in aspartate transaminase (AST) | Baseline to 6 months
  Relative change (%) in AST at 6 months (T1) from baseline (T0).
Change in alkaline phosphatase (ALP) | Baseline to 6 months
  Relative change (%) in ALP at 6 months (T1) from baseline (T0).
Change in c-reactive protein (CRP) | Baseline to 6 months
  Relative change (%) in CRP at 6 months (T1) from baseline (T0).
Change in Fibrosis-4 Index (FIB-4) | Baseline to 6 months
  Relative change (%) in FIB-4 at 6 months (T1) from baseline (T0).
Change in Enhanced Liver Fibrosis test (ELF) | Baseline to 6 months
  Relative change (%) in ELF at 6 months (T1) from baseline (T0).
Change in Nonalcoholic steatohepatitis related biomarkers score (NIS4) | Baseline to 6 months
  Relative change (%) in NIS4 at 6 months (T1) from baseline (T0).
Change in liver stiffness | Baseline to 6 months
  Relative change (%) in liver stiffness as measured by transient elastography at 6 months (T1) from baseline (T0).
Change in hepatic fat deposition | Baseline to 6 months
  Relative change (%) in hepatic fat deposition as measured by magnetic resonance imaging (MRI) with proton density fat fraction (PDFF) at 6 months (T1) from baseline (T0).

SECONDARY OUTCOMES:
Change in total body weight | Baseline to 12 months
  Relative change (%) in total body weight at 1 year (T2) from 6 months (T1) and baseline (T0).
Change in bilirubin | Baseline to 12 months
  Relative change (%) in bilirubin at 1 year (T2) from 6 months (T1) and baseline (T0).
Change in alanine transaminase (ALT) | Baseline to 12 months
  Relative change (%) in ALT at 1 year (T2) from 6 months (T1) and baseline (T0).
Change in aspartate transaminase (AST) | Baseline to 12 months
  Relative change (%) in AST at 1 year (T2) from 6 months (T1) and baseline (T0).
Change in c-reactive protein (CRP) | Baseline to 12 months
  Relative change (%) in CRP at 1 year (T2) from 6 months (T1) and baseline (T0).
Change in Fibrosis-4 Index (FIB-4) | Baseline to 12 months
  Relative change (%) in FIB-4 at 1 year (T2) from 6 months (T1) and baseline (T0).
Change in Enhanced Liver Fibrosis test (ELF) | Baseline to 12 months
  Relative change (%) in ELF at 1 year (T2) from 6 months (T1) and baseline (T0).
Change in Nonalcoholic steatohepatitis related biomarkers score (NIS4) | Baseline to 12 months
  Relative change (%) in NIS4 at 1 year (T2) from 6 months (T1) and baseline (T0).
Change in alkaline phosphatase (ALP) | Baseline to 12 months
  Relative change (%) in ALP at 1 year (T2) from 6 months (T1) and baseline (T0).
Change in hepatic fat deposition | Baseline to 12 months
  Relative change (%) in hepatic fat deposition as measured by magnetic resonance imaging (MRI) with proton density fat fraction (PDFF) at 1 year (T2) from 6 months (T1) and baseline (T0).

CONTACTS AND LOCATIONS:
Overall Officials: Arun J Sanyal, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No